CLINICAL TRIAL: NCT03343496
Title: Simplification and Implementation of Awake Fibreoptic Orotracheal Intubation
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Shengjin Ge,MD, Professor of Anesthesiology, Fudan University
Other Study IDs: B2017-112R
Record Dates: First submitted 2017-11-11; First posted 2017-11-17 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; Trachea; Intubation
Keywords: Awake fiberoptic intubation
MeSH Terms: conditions — Tracheal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Awake fiberoptic intubation (AFOI) — With forty patients (ASA I~II, aged 18~75, simulating cervical instability injury) recruited to be operated on under general anesthesia, two experienced anesthesiologists performed the whole procedures within the study. Pre anesthetic interview was taken to illustrate the procedures of tracheal intubation to the patients. The simplified method consisted of three parts: conscious sedation, regional anesthesia and intubation. The time of AFOI, rate of one-time intubation success, hemodynamic parameters, pulse oxygen saturation (SpO2), rate of amnesia of the intubation, patients' satisfaction, and relative complications were recorded accordingly.

SUMMARY:
Awake fibreoptic intubation (AFOI) is a classic and standard method for some special patients which is also difficult for anesthesiologists to learn and master. The procedure is sometimes hard and often takes about 20-30 min. Most of patients have a strong sense of discomfort. Investigators conducted the research to study the simplification and feasibility of AFOI.

DETAILED DESCRIPTION:
Many studies have studied the sedative drugs and regional anesthesia related to awake intubation. However, several problems of AFOI are existing including long operation time, patients' strong discomfort, coughing and resistance. And, to investigators' knowledge, there was a lack of a fixed procedure for the implementation of AFOI. Investigators conducted the research and aimed to study the simplification and feasibility of a new AFOI method based on years of clinical theory, practice and experience.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists' physical status I-II patients
2. Aged 18-75 years
3. Mallampati Grade I-II
4. Body Mass Index 18.5-28 kg·m-2

Exclusion Criteria:

1. Allergic to the drugs involved in the study
2. Neck mass or infection
3. Drug or alcohol abuse
4. Pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The trial will be performed at Zhongshan Hospital, Fudan University in Shanghai, China.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
The average total time of Awake Fiberoptic Orotracheal Intubation (AFOI) | End of the AFOI
  The time from the midazolam injection to positive end tidal CO2 acquired (Minutes)
The rate of one-time intubation success. | End of the AFOI
  All steps are successful once (Percentage)

SECONDARY OUTCOMES:
Systolic blood pressure, SBP (mmHg) | During the AFOI
  SBP is used to assess hemodynamic fluctuations
Diastolic blood pressure, DBP (mmHg) | During the AFOI
  DBP is used to assess hemodynamic fluctuations
Heart rate, HR (bpm) | During the AFOI
  HR is used to assess hemodynamic fluctuations
Rate of amnesia of the intubation | On the first postoperative day
  It is used to assess anterograde amnesia of midazolam
Ramsay sedation scale | During the AFOI
  1= anxious or restless or both, 2 = cooperative, orientated and tranquil, 3 = responding to commands, 4 = brisk response to stimulus, 5 = sluggish response to stimulus, 6= No response to stimulus
Patients' satisfaction | On the first postoperative day
  1 = excellent, 2 = good, 3 = fair, 4 = poor
Unexpected coughing | During the AFOI
  Unexpected coughing was evaluated with 4 score (1=none, 2< 3 times unexpected slight coughing comparable to 'clearing ones' throat', 3≥2 times, mild unexpected coughing lasting less than a minute, 4=persistent unexpected coughing)
Relative complications | End of the surgery and the first postoperative day
  Such as arrhythmias, bleeding or sore throat
Vocal cord movement | During the AFOI
  1 = open, 2 = moving, 3 = closing, 4 = closed
Hypoxic episode | During the AFOI
  SpO2<90%

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided